CLINICAL TRIAL: NCT02785237
Title: Intra-patient Randomized Study With Polymer Free Drug Eluting Stent Versus Abluminal Biodegradable Polymer Drug Eluting Stent With Early OCT Follow up
Brief Title: Intra-patient Study With Polymer Free Drug Eluting Stent Versus Abluminal Biodegradable Polymer Drug Eluting Stent With Early OCT (Optical Coherence Tomography) Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRIENDLY OCT
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stent; OCT; Re-endothelialization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Coroflex® ISAR Drug-eluting stent in first lesion (Active Comparator): Patients with Coroflex® ISAR Drug-eluting stent in the first lesion
  Interventions: Device: Coroflex® ISAR Drug-eluting stent
- Ultimaster® Drug-eluting stent in first lesion (Active Comparator): Patients with Ultimaster® Drug-eluting stent in first lesion
  Interventions: Device: Ultimaster® Drug-eluting stent
- Coroflex® ISAR Drug-eluting stent in second lesion (Active Comparator): Patients with with Ultimaster® Drug-eluting stent in first lesion
  Interventions: Device: Coroflex® ISAR Drug-eluting stent
- Ultimaster® Drug-eluting stent in second lesion (Active Comparator): Patients with Coroflex® ISAR Drug-eluting stent in the first lesion
  Interventions: Device: Ultimaster® Drug-eluting stent

INTERVENTIONS:
Device: Coroflex® ISAR Drug-eluting stent — Coroflex® ISAR Drug-eluting stent and an Ultimaster® Drug-eluting stent in the second lesion.
  Arms: Coroflex® ISAR Drug-eluting stent in first lesion; Coroflex® ISAR Drug-eluting stent in second lesion
Device: Ultimaster® Drug-eluting stent — Ultimaster® Drug-eluting stent and a Coroflex® ISAR Drug-eluting stent in the second lesion.
  Arms: Ultimaster® Drug-eluting stent in first lesion; Ultimaster® Drug-eluting stent in second lesion

SUMMARY:
The objective of the study is to evaluate the process of early re-endothelialization of the Coroflex® ISAR Drug-eluting stent compared with the Ultimaster® Drug-eluting stent

DETAILED DESCRIPTION:
The objective of the study is to evaluate the process of early re-endothelialization of the Coroflex® ISAR Drug-eluting stent compared with the Ultimaster® Drug-eluting stent

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Signature of informed consent
* Patients with angina and a clinical indication for coronary revascularisation with a drug-eluting stent
* Presence of at least 2 lesions to be revascularised with similar angiographic characteristics

  * Reference lesion diameter with at most a difference of 0.5 mm
  * Maximum difference in lesion length of 10 mm
  * Lesions able to be treated with only 1 stent

Exclusion Criteria:

* Lesions due to restenosis
* Lesions in saphenous vein grafts
* STE-ACS ( ST elevation- Acute Coronary Syndrome)
* Cardiogenic shock
* Dual antiplatelet therapy contraindication for> 3 months
* Follow-up catheterisation contraindicated

  * Chronic kidney failure with creatinine > 2 mg/dL
  * Allergy to iodinated contrast agents
  * Serious complication from vascular access in previous catheterisation
* Ineligible for evaluation via optical coherence tomography

  * Lesion located <5 mm from aorto-ostial junction
  * Severe proximal angulation >90º
* Bifurcation lesion requiring a strategy with two stents
* Angiographic characteristics that promote stent malposition

  * Aneurysm or coronary artery ectasia
  * Presence of a thrombus classed as TIMI (Thrombolysis In Myocardial Infarction )2 flow or higher
  * Severe calcification, in particular in cases of calcium spike
  * Severe lesion angulation
* Inability to do reliable follow-up, in the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of early coating on the struts of the Coroflex® ISAR Drug-eluting stent versus Ultimaster® - Drug eluting stent at 3 months OCT after stent implantation. | 3 months
Percentage of covered struts at 3 months OCT after stent implantation. | 3 months
Percentage of stents with ≥3% of uncovered struts at 3 months OCT after stent implantation. | 3 months
Percentage of uncovered struts ≥3% at 3 months OCT after stent implantation. | 3 months
Number of transversal sections with a percentage (rate of uncovered struts/ total number of struts) > 30 % at 3 months OCT after stent implantation. | 3 months

SECONDARY OUTCOMES:
Percentage of covered struts, at 1 month, 2 months and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Total Tissue coverage at 1month, 2 months and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Mean thickness of struts tissue coverage at 1 month, 2 months and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
MACE (Major Adverse Cardiac Events) at 30 days, 3 months, 6 months and 12 months. | 30 days and 3 months and 6 months and 12 months
Target lesion revascularization and target vessel revascularization at 30 days, 3 months, 6 months and 12 months OCT after stent implantation . | 30 days and 3 months and 6 months and 12 months
Percentage of stent malapposition at 1 month and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Percentage of struts malapposition at 1 month and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Percentage of struts malapposition> 260 µm at 1 month and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Percentage of stents with any malapposition strut > 260 µm at 1 month and 3 months OCT after stent implantation. | 1 month and 2 months and 3 months
Healing Score at 1 month and 3 months OCT after stent implantation . | 1 month and 2 months and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno García del Blanco, MD, PhD, Study Director — Hospital Universitari Vall d'Hebron (Barcelona)
Locations (3):
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de León, León

REFERENCES:
- [Background] Stone GW, Moses JW, Ellis SG, Schofer J, Dawkins KD, Morice MC, Colombo A, Schampaert E, Grube E, Kirtane AJ, Cutlip DE, Fahy M, Pocock SJ, Mehran R, Leon MB. Safety and efficacy of sirolimus- and paclitaxel-eluting coronary stents. N Engl J Med. 2007 Mar 8;356(10):998-1008. doi: 10.1056/NEJMoa067193. Epub 2007 Feb 12. PMID 17296824
- [Background] Kirtane AJ, Gupta A, Iyengar S, Moses JW, Leon MB, Applegate R, Brodie B, Hannan E, Harjai K, Jensen LO, Park SJ, Perry R, Racz M, Saia F, Tu JV, Waksman R, Lansky AJ, Mehran R, Stone GW. Safety and efficacy of drug-eluting and bare metal stents: comprehensive meta-analysis of randomized trials and observational studies. Circulation. 2009 Jun 30;119(25):3198-206. doi: 10.1161/CIRCULATIONAHA.108.826479. Epub 2009 Jun 15. PMID 19528338
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] de la Torre-Hernandez JM, Alfonso F, Hernandez F, Elizaga J, Sanmartin M, Pinar E, Lozano I, Vazquez JM, Botas J, Perez de Prado A, Hernandez JM, Sanchis J, Nodar JM, Gomez-Jaume A, Larman M, Diarte JA, Rodriguez-Collado J, Rumoroso JR, Lopez-Minguez JR, Mauri J; ESTROFA Study Group. Drug-eluting stent thrombosis: results from the multicenter Spanish registry ESTROFA (Estudio ESpanol sobre TROmbosis de stents FArmacoactivos). J Am Coll Cardiol. 2008 Mar 11;51(10):986-90. doi: 10.1016/j.jacc.2007.10.057. PMID 18325436
- [Background] Kolh P, Windecker S, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; European Society of Cardiology Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; EACTS Clinical Guidelines Committee; Sousa Uva M, Achenbach S, Pepper J, Anyanwu A, Badimon L, Bauersachs J, Baumbach A, Beygui F, Bonaros N, De Carlo M, Deaton C, Dobrev D, Dunning J, Eeckhout E, Gielen S, Hasdai D, Kirchhof P, Luckraz H, Mahrholdt H, Montalescot G, Paparella D, Rastan AJ, Sanmartin M, Sergeant P, Silber S, Tamargo J, ten Berg J, Thiele H, van Geuns RJ, Wagner HO, Wassmann S, Wendler O, Zamorano JL; Task Force on Myocardial Revascularization of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery; European Association of Percutaneous Cardiovascular Interventions. 2014 ESC/EACTS Guidelines on myocardial revascularization: the Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2014 Oct;46(4):517-92. doi: 10.1093/ejcts/ezu366. Epub 2014 Aug 29. No abstract available. PMID 25173601
- [Background] Ferreira-Gonzalez I, Marsal JR, Ribera A, Permanyer-Miralda G, Garcia-Del Blanco B, Marti G, Cascant P, Martin-Yuste V, Brugaletta S, Sabate M, Alfonso F, Capote ML, De La Torre JM, Ruiz-Lera M, Sanmiguel D, Cardenas M, Pujol B, Baz JA, Iniguez A, Trillo R, Gonzalez-Bejar O, Casanova J, Sanchez-Gila J, Garcia-Dorado D. Background, incidence, and predictors of antiplatelet therapy discontinuation during the first year after drug-eluting stent implantation. Circulation. 2010 Sep 7;122(10):1017-25. doi: 10.1161/CIRCULATIONAHA.110.938290. Epub 2010 Aug 23. PMID 20733100
- [Background] D'Ascenzo F, Bollati M, Clementi F, Castagno D, Lagerqvist B, de la Torre Hernandez JM, ten Berg JM, Brodie BR, Urban P, Jensen LO, Sardi G, Waksman R, Lasala JM, Schulz S, Stone GW, Airoldi F, Colombo A, Lemesle G, Applegate RJ, Buonamici P, Kirtane AJ, Undas A, Sheiban I, Gaita F, Sangiorgi G, Modena MG, Frati G, Biondi-Zoccai G. Incidence and predictors of coronary stent thrombosis: evidence from an international collaborative meta-analysis including 30 studies, 221,066 patients, and 4276 thromboses. Int J Cardiol. 2013 Jul 31;167(2):575-84. doi: 10.1016/j.ijcard.2012.01.080. Epub 2012 Feb 22. PMID 22360945
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Background] Hassan AK, Bergheanu SC, Stijnen T, van der Hoeven BL, Snoep JD, Plevier JW, Schalij MJ, Wouter Jukema J. Late stent malapposition risk is higher after drug-eluting stent compared with bare-metal stent implantation and associates with late stent thrombosis. Eur Heart J. 2010 May;31(10):1172-80. doi: 10.1093/eurheartj/ehn553. Epub 2009 Jan 21. PMID 19158118
- [Background] Lee CW, Kang SJ, Park DW, Lee SH, Kim YH, Kim JJ, Park SW, Mintz GS, Park SJ. Intravascular ultrasound findings in patients with very late stent thrombosis after either drug-eluting or bare-metal stent implantation. J Am Coll Cardiol. 2010 May 4;55(18):1936-42. doi: 10.1016/j.jacc.2009.10.077. PMID 20430265
- [Background] Alfonso F, Dutary J, Paulo M, Gonzalo N, Perez-Vizcayno MJ, Jimenez-Quevedo P, Escaned J, Banuelos C, Hernandez R, Macaya C. Combined use of optical coherence tomography and intravascular ultrasound imaging in patients undergoing coronary interventions for stent thrombosis. Heart. 2012 Aug;98(16):1213-20. doi: 10.1136/heartjnl-2012-302183. PMID 22826559
- [Background] Guagliumi G, Sirbu V, Musumeci G, Gerber R, Biondi-Zoccai G, Ikejima H, Ladich E, Lortkipanidze N, Matiashvili A, Valsecchi O, Virmani R, Stone GW. Examination of the in vivo mechanisms of late drug-eluting stent thrombosis: findings from optical coherence tomography and intravascular ultrasound imaging. JACC Cardiovasc Interv. 2012 Jan;5(1):12-20. doi: 10.1016/j.jcin.2011.09.018. PMID 22230145
- [Background] Cook S, Ladich E, Nakazawa G, Eshtehardi P, Neidhart M, Vogel R, Togni M, Wenaweser P, Billinger M, Seiler C, Gay S, Meier B, Pichler WJ, Juni P, Virmani R, Windecker S. Correlation of intravascular ultrasound findings with histopathological analysis of thrombus aspirates in patients with very late drug-eluting stent thrombosis. Circulation. 2009 Aug 4;120(5):391-9. doi: 10.1161/CIRCULATIONAHA.109.854398. Epub 2009 Jul 20. PMID 19620501
- [Background] Kolandaivelu K, Swaminathan R, Gibson WJ, Kolachalama VB, Nguyen-Ehrenreich KL, Giddings VL, Coleman L, Wong GK, Edelman ER. Stent thrombogenicity early in high-risk interventional settings is driven by stent design and deployment and protected by polymer-drug coatings. Circulation. 2011 Apr 5;123(13):1400-9. doi: 10.1161/CIRCULATIONAHA.110.003210. Epub 2011 Mar 21. PMID 21422389
- [Background] Palmerini T, Biondi-Zoccai G, Della Riva D, Stettler C, Sangiorgi D, D'Ascenzo F, Kimura T, Briguori C, Sabate M, Kim HS, De Waha A, Kedhi E, Smits PC, Kaiser C, Sardella G, Marullo A, Kirtane AJ, Leon MB, Stone GW. Stent thrombosis with drug-eluting and bare-metal stents: evidence from a comprehensive network meta-analysis. Lancet. 2012 Apr 14;379(9824):1393-402. doi: 10.1016/S0140-6736(12)60324-9. Epub 2012 Mar 23. PMID 22445239
- [Background] Raber L, Magro M, Stefanini GG, Kalesan B, van Domburg RT, Onuma Y, Wenaweser P, Daemen J, Meier B, Juni P, Serruys PW, Windecker S. Very late coronary stent thrombosis of a newer-generation everolimus-eluting stent compared with early-generation drug-eluting stents: a prospective cohort study. Circulation. 2012 Mar 6;125(9):1110-21. doi: 10.1161/CIRCULATIONAHA.111.058560. Epub 2012 Feb 1. PMID 22302840
- [Background] de la Torre Hernandez JM, Alfonso F, Gimeno F, Diarte JA, Lopez-Palop R, Perez de Prado A, Rivero F, Sanchis J, Larman M, Diaz JF, Elizaga J, Moreiras JM, Gomez Jaume A, Hernandez JM, Mauri J, Recalde AS, Bullones JA, Rumoroso JR, Del Blanco BG, Baz JA, Bosa F, Botas J, Hernandez F; ESTROFA-2 Study Group. Thrombosis of second-generation drug-eluting stents in real practice results from the multicenter Spanish registry ESTROFA-2 (Estudio Espanol Sobre Trombosis de Stents Farmacoactivos de Segunda Generacion-2). JACC Cardiovasc Interv. 2010 Sep;3(9):911-9. doi: 10.1016/j.jcin.2010.06.010. PMID 20850089
- [Background] Bangalore S, Kumar S, Fusaro M, Amoroso N, Attubato MJ, Feit F, Bhatt DL, Slater J. Short- and long-term outcomes with drug-eluting and bare-metal coronary stents: a mixed-treatment comparison analysis of 117 762 patient-years of follow-up from randomized trials. Circulation. 2012 Jun 12;125(23):2873-91. doi: 10.1161/CIRCULATIONAHA.112.097014. Epub 2012 May 14. PMID 22586281
- [Background] Sarno G, Lagerqvist B, Frobert O, Nilsson J, Olivecrona G, Omerovic E, Saleh N, Venetzanos D, James S. Lower risk of stent thrombosis and restenosis with unrestricted use of 'new-generation' drug-eluting stents: a report from the nationwide Swedish Coronary Angiography and Angioplasty Registry (SCAAR). Eur Heart J. 2012 Mar;33(5):606-13. doi: 10.1093/eurheartj/ehr479. Epub 2012 Jan 9. PMID 22232428
- [Background] de la Torre Hernandez JM. Late acquired incomplete stent apposition: incidence, mechanisms and clinical implications. EuroIntervention. 2009 May;5 Suppl D:D112-20. PMID 19736059
- [Background] Schulz S, Schuster T, Mehilli J, Byrne RA, Ellert J, Massberg S, Goedel J, Bruskina O, Ulm K, Schomig A, Kastrati A. Stent thrombosis after drug-eluting stent implantation: incidence, timing, and relation to discontinuation of clopidogrel therapy over a 4-year period. Eur Heart J. 2009 Nov;30(22):2714-21. doi: 10.1093/eurheartj/ehp275. Epub 2009 Jul 11. PMID 19596658
- [Background] Airoldi F, Colombo A, Morici N, Latib A, Cosgrave J, Buellesfeld L, Bonizzoni E, Carlino M, Gerckens U, Godino C, Melzi G, Michev I, Montorfano M, Sangiorgi GM, Qasim A, Chieffo A, Briguori C, Grube E. Incidence and predictors of drug-eluting stent thrombosis during and after discontinuation of thienopyridine treatment. Circulation. 2007 Aug 14;116(7):745-54. doi: 10.1161/CIRCULATIONAHA.106.686048. Epub 2007 Jul 30. PMID 17664375
- [Background] Valgimigli M, Campo G, Monti M, Vranckx P, Percoco G, Tumscitz C, Castriota F, Colombo F, Tebaldi M, Fuca G, Kubbajeh M, Cangiano E, Minarelli M, Scalone A, Cavazza C, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R; Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia Study (PRODIGY) Investigators. Short- versus long-term duration of dual-antiplatelet therapy after coronary stenting: a randomized multicenter trial. Circulation. 2012 Apr 24;125(16):2015-26. doi: 10.1161/CIRCULATIONAHA.111.071589. Epub 2012 Mar 21. PMID 22438530
- [Background] Gwon HC, Hahn JY, Park KW, Song YB, Chae IH, Lim DS, Han KR, Choi JH, Choi SH, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Jang Y, Kim HS. Six-month versus 12-month dual antiplatelet therapy after implantation of drug-eluting stents: the Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting (EXCELLENT) randomized, multicenter study. Circulation. 2012 Jan 24;125(3):505-13. doi: 10.1161/CIRCULATIONAHA.111.059022. Epub 2011 Dec 16. PMID 22179532
- [Background] Kim BK, Hong MK, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Kang TS, Park BE, Kang WC, Lee SH, Yoon JH, Hong BK, Kwon HM, Jang Y; RESET Investigators. A new strategy for discontinuation of dual antiplatelet therapy: the RESET Trial (REal Safety and Efficacy of 3-month dual antiplatelet Therapy following Endeavor zotarolimus-eluting stent implantation). J Am Coll Cardiol. 2012 Oct 9;60(15):1340-8. doi: 10.1016/j.jacc.2012.06.043. Epub 2012 Sep 19. PMID 22999717
- [Background] Cassese S, Byrne RA, Tada T, King LA, Kastrati A. Clinical impact of extended dual antiplatelet therapy after percutaneous coronary interventions in the drug-eluting stent era: a meta-analysis of randomized trials. Eur Heart J. 2012 Dec;33(24):3078-87. doi: 10.1093/eurheartj/ehs318. Epub 2012 Oct 22. PMID 23091199
- [Background] Navarese EP, Kubica J, Castriota F, Gibson CM, De Luca G, Buffon A, Bolognese L, Margheri M, Andreotti F, Di Mario C, De Servi S. Safety and efficacy of biodegradable vs. durable polymer drug-eluting stents: evidence from a meta-analysis of randomised trials. EuroIntervention. 2011 Dec;7(8):985-94. doi: 10.4244/EIJV7I8A155. PMID 22116195
- [Background] Stefanini GG, Byrne RA, Serruys PW, de Waha A, Meier B, Massberg S, Juni P, Schomig A, Windecker S, Kastrati A. Biodegradable polymer drug-eluting stents reduce the risk of stent thrombosis at 4 years in patients undergoing percutaneous coronary intervention: a pooled analysis of individual patient data from the ISAR-TEST 3, ISAR-TEST 4, and LEADERS randomized trials. Eur Heart J. 2012 May;33(10):1214-22. doi: 10.1093/eurheartj/ehs086. Epub 2012 Mar 24. PMID 22447805
- [Background] Zhong JK, Guo ZG, Li C, Wang ZK, Lai WY, Tu Y. Probucol alleviates atherosclerosis and improves high density lipoprotein function. Lipids Health Dis. 2011 Nov 12;10:210. doi: 10.1186/1476-511X-10-210. PMID 22078494
- [Background] Guo YS, Wang CX, Cao J, Gao JL, Zou X, Ren YH, Fan L. Antioxidant and lipid-regulating effects of probucol combined with atorvastatin in patients with acute coronary syndrome. J Thorac Dis. 2015 Mar;7(3):368-75. doi: 10.3978/j.issn.2072-1439.2014.12.29. PMID 25922714
- [Background] Smits PC, Chevalier B. DISCOVERY 1TO3 polymer DES at 1 , 2 and 3 months after stent. 2(1).
- [Background] Raber L, Onuma Y, Brugaletta S, Garcia-Garcia HM, Backx B, Iniguez A, Okkels Jensen L, Cequier-Fillat A, Pilgrim T, Christiansen EH, Hofma SH, Suttorp M, Serruys PW, Sabate M, Windecker S. Arterial healing following primary PCI using the Absorb everolimus-eluting bioresorbable vascular scaffold (Absorb BVS) versus the durable polymer everolimus-eluting metallic stent (XIENCE) in patients with acute ST-elevation myocardial infarction: rationale and design of the randomised TROFI II study. EuroIntervention. 2016 Jul 20;12(4):482-9. doi: 10.4244/EIJY15M08_03. PMID 26342471
- [Derived] Otaegui Irurueta I, Gonzalez Sucarrats S, Barron Molina JL, Perez de Prado A, Massotti M, Carmona Ramirez MA, Marti G, Bellera N, Serra B, Serra V, Domingo E, Lopez-Benito M, Sabate M, Ferreira Gonzalez I, Garcia Del Blanco B. Can an ultrathin strut stent design and a polymer free, proendothelializing probucol matrix coating improve early strut healing? The FRIENDLY-OCT trial. An intra-patient randomized study with OCT, evaluating early strut coverage of a novel probucol coated polymer-free and ultra-thin strut sirolimus-eluting stent compared to a biodegradable polymer sirolimus-eluting stent. Int J Cardiol. 2022 Aug 1;360:13-20. doi: 10.1016/j.ijcard.2022.04.043. Epub 2022 Apr 25. PMID 35472561